CLINICAL TRIAL: NCT02221557
Title: Clinical and Histomorphometric Evaluation of Beta-tricalcium Phosphate/Polylactide Bone Substitute for Socket Preservation
Brief Title: Case Series of New Alloplastic Bone Graft Material
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunstar Americas (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-7-1-1
Record Dates: First submitted 2014-08-14; First posted 2014-08-20 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-07

CONDITIONS: Periodontology; Oral Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- New alloplastic bone graft material (Experimental)
  Interventions: Device: easy-graft (beta-Tricalcium Phosphate)

INTERVENTIONS:
Device: easy-graft (beta-Tricalcium Phosphate)

SUMMARY:
A case series to compare the handling and effectiveness of two different treatment approaches using a new alloplastic bone graft material in ridge preservation compared to allograft existing historical data.

ELIGIBILITY:
Inclusion Criteria:

* Must have read, understood and signed a consent form.
* 18-75 years of age
* Diagnosis with a need of extraction of single tooth (with intact extraction socket at the time of extraction) with adjacent teeth present.

Exclusion Criteria:

* Active caries or endodontic lesions in adjacent teeth
* Any systemic disease or condition that would compromise the normal healing. (e.g., uncontrolled diabetes)
* Taking any medication known for gingival hyperplasia for past 3 months.
* Any systemic contraindications to surgery
* Subject smokes > 10 cigarettes per day.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Dentistry, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- New Alloplastic Bone Graft Material: easy-graft (beta-Tricalcium Phosphate)
Period: Overall Study
Arm/Group | New Alloplastic Bone Graft Material
Started | 8
Completed | 5
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | New Alloplastic Bone Graft Material
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Widest ridge width [Mean (Standard Deviation); unit: mm] | 9.3 (2.5)
Deepest vertical depth [Mean (Standard Deviation); unit: mm] | 10.0 (2.3)
Widest open [Mean (Standard Deviation); unit: mm] | 8.3 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Radiographic Measurement of Alveolar Ridge Height
Description: Radiographic measurement was taken at most-middle portion of the grafted site, perpendicular to the line drawn from reference point (e.g. adjacent tooth/teeth Cement-Enamel Junction (CEJ) or margin of the restoration).
Time Frame: Change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | New Alloplastic Bone Graft Material
Number analyzed (Participants) | 5
percentage of change | 1.2 (6.2)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | New Alloplastic Bone Graft Material
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is at least 30 days from the time submitted to the sponsor for review. Sponsor reserves the right to require the PI to remove sponsor's confidential information. Upon sponsor's written request, publication will be delayed up to 60 days to enable sponsor to secure adequate intellectual property protection.